CLINICAL TRIAL: NCT03095482
Title: tDCS-Augmented Exposure Therapy for Pathological Fear
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Michael J. Telch, Professor of Psychology, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2016-02-0024
Record Dates: First submitted 2017-03-20; First posted 2017-03-29 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Specific Phobias
Keywords: Arachnophobia (fear of spiders); Ophidophobia (fear of snakes); Germaphobia (fear of germs, dirtiness, and contamination)
MeSH Terms: conditions — Phobia, Specific; Arachnophobia; Zoophobia; Mysophobia | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to receive either (a) excitatory tDCS of the medial prefrontal cortex and inhibitory tDCS of right dorsolateral prefrontal cortex, or (b) sham tDCS
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, treatment administrators, and outcome assessors will be blind to tDCS condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tDCS + In Vivo Exposure (Active Comparator): Participants assigned to this condition will receive excitatory transcranial direct current stimulation (tDCS) of the left medial prefrontal cortex (lmPFC) and inhibitory tDCS of right dorsolateral prefrontal cortex (rdlPFC). tDCS will be administered for 20 minutes at 1.7 mA, followed by 30 minutes of in vivo exposure therapy.
  Interventions: Device: Transcranial Direct Current Stimulation (tDCS); Behavioral: In vivo exposure therapy
- sham tDCS + In Vivo Exposure (Sham Comparator): Participants assigned to this condition will receive sham transcranial direct current stimulation (tDCS), which will consist of 30 seconds of stimulation at the beginning and end of tDCS administration. Electrode positioning will be counterbalanced across participants (i.e., either mPFC+ or mPFC-, with same electrode positioning as the active comparators). Sham tDCS will be administered for 20 minutes, followed by 30 minutes of in vivo exposure therapy.
  Interventions: Behavioral: In vivo exposure therapy

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation (tDCS) — Participants will receive 20 minutes of either active or sham tDCS prior to in vivo exposure to feared targets.
  Arms: Active tDCS + In Vivo Exposure
Behavioral: In vivo exposure therapy — Participants will receive 30 minutes of in vivo exposure to feared targets following either active or sham tDCS

SUMMARY:
This double-blind randomized controlled clinical trial aims to test whether transcranial direct current stimulation (tDCS) can be used to modulate fear extinction learning during exposure therapy for pathological fear, including fear of spiders, snakes, or germs / contamination. Participation takes place over three laboratory visits, including (1) a pre-treatment visit, (2) a treatment and post-treatment visit, and (3) a 1 month follow-up visit. During treatment, participants will receive either 20 minutes of active or sham tDCS, followed by 30 minutes of in vivo exposure therapy.

DETAILED DESCRIPTION:
In a trans-diagnostic sample with marked pathological fear and behavioral avoidance, this study aims to: (1) evaluate whether excitatory tDCS of the mPFC and inhibitory tDCS of right dlPFC enhances exposure therapy relative to sham tDCS; (2) determine whether tDCS effects are moderated by baseline negative prognostic indicators; and (3) determine whether tDCS effects are mediated by pre-post changes in vigilance to threat, in-session fear reduction, and contextual memory for the exposure context. If successful, the project may discover a potentially effective exposure therapy augmentation, and may enhance knowledge of the behavioral, cognitive, affective, and neurobiological factors that moderate and mediate acute treatment response and maintenance of treatment gains. This knowledge may inform treatment development efforts for more debilitating forms of pathological fear.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65.
2. Fluent in English.
3. A score on at least 1 fear domain-specific prescreen measure > 2 SDs above the subject pool prescreen mean. These measures include (a) FSQ, and (b) OCI-R.
4. Peak fear ≥ 50 on BATs 1 and 2.

Exclusion Criteria:

1. Currently receiving treatment for the primary fear domain (based on clinical interview).
2. Unstable dose of psychotropic medications within 6 weeks prior to baseline assessment (based on the DMQ; see measures).
3. Medical condition that would contraindicate participation in treatment or assessment activities (e.g., cardiovascular problems; based on the DMQ; see measures).
4. Pregnancy (based on the DMQ; see measures).
5. Current major depressive disorder (based on MINI; see measures).
6. Current, or history of bipolar disorder (based on MINI; see measures).
7. Current, or history of psychotic symptoms (based on MINI; see measures).
8. Serious suicidal risk, as determined by self-report (C-SSRS, BDI-II) and clinical interview (MINI; see measures).
9. Active neurological conditions, including seizures, stroke, unexplained loss of consciousness or concussion (based on DMQ and tDCS Safety Screening Form; see measures)
10. Contraindications for tDCS: Metal in the head or implanted brain medical devices.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-09-06 (Actual); Study Completion 2018-09-06 (Actual)

PRIMARY OUTCOMES:
Change in peak fear during two behavioral approach tasks across time-points. | Pre-treatment (baseline), post-treatment (1 week later), and follow-up (1 month after treatment)
  Subjective units of distress from 0 = no fear, to 100 = extreme fear
Change in approach level during two behavioral approach tasks across time points. | Pre-treatment (baseline), post-treatment (1 week later), and follow-up (1 month after treatment)
  Highest difficulty level achieved from 0 = least challenging to 10 = most challenging.

SECONDARY OUTCOMES:
Change in arachnophobia symptom severity across time-points | Pre-treatment (baseline), post-treatment (1 week later), and follow-up (1 month after treatment)
  Total score on the Fear of Spiders Questionnaire
Change in ophidophobia symptom severity across time-points | Pre-treatment (baseline), post-treatment (1 week later), and follow-up (1 month after treatment)
  Total score on the Fear of Snakes Questionnaire
Change in germaphobia / contamination fear symptom severity across time points. | Pre-treatment (baseline), post-treatment (1 week later), and follow-up (1 month after treatment)
  Total score on the Obsessive Compulsive Inventory - Revised.
Threat vigilance task | Before and after tDCS administration (1 week after baseline)
  Computer-based task that assesses attention biases towards and away from threatening images.
Visuospatial working memory task | Before and after tDCS administration (1 week after baseline)
  Delayed match to sample task assessing recognition of 4 x 4 arrays of colored blocks, after a brief delay.
Incidental contextual memory task | Stimulus presented during in vivo exposure (1 week after baseline), and memory assessed at follow-up (1 month after treatment)
  Assessment of incidental memory for a 4 x 4 array of line drawings from the Test of Memory Malingering, presented in the treatment context only during in vivo exposure.

CONTACTS AND LOCATIONS:
Overall Officials: Adam R. Cobb, Ph.D., Principal Investigator — The University of Texas at Austin; Michael J. Telch, PhD, Study Director — The University of Texas at Austin
Locations (1):
- Laboratory for the Study of Anxiety Disorders, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Website for the Laboratory for the Study of Anxiety Disorders — http://UTanxiety.com